CLINICAL TRIAL: NCT00259337
Title: Immunogenicity and Safety of the Sanofi Pasteur DTacP-IPV//PRP~T Combined Vaccine (PENTAXIM™) Given as a Three-Dose Primary Vaccination at 6, 10, and 14 Weeks of Age and Followed by a Booster Dose at 18-19 Months of Age in Healthy Infants in India.
Brief Title: Immunogenicity and Safety of Pentaxim™ in an Indian Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2I41
Record Dates: First submitted 2005-11-24; First posted 2005-11-29 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Diphtheria; Tetanus; Polio; Pertussis; Haemophilus Infections
Keywords: Diphteria; Tetanus; Polio; Acellular Pertussis; Hib; Haemophilus influenzae type B
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis; Whooping Cough; Haemophilus Infections | interventions — Pentavac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Diphteria/Tetanus/Polio/Acellular Pertussis/Hib vaccine

INTERVENTIONS:
Biological: Diphteria/Tetanus/Polio/Acellular Pertussis/Hib vaccine — 0.5 mL, IM
  Other Names: PENTAXIM™

SUMMARY:
The present clinical study will assess the immunogenicity as the primary objective and the reactogenicity as the secondary objective of Aventis Pasteur's DTacP-IPV// PRP~T combined vaccine (Pentavac™ or Pentaxim™) as a three-dose primary vaccination at 6, 10 and 14 weeks of age followed by a booster dose during the second year of life.

Safety:

This study will describe the safety after each dose of the primary series of the study's combined vaccine (Pentaxim™).

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 56 days inclusive on the day of inclusion
* Born at full term pregnancy (> 37 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the (first) trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past.
* Any vaccination preceding the trial vaccination (except BCG and hepatitis B)
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B or Haemophilus influenza type b (confirmed either clinically, serologically or microbiologically).
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis diseases or Haemophilus influenza type b infection with the trial vaccine or another vaccine.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current seizures
* Febrile illness (rectal temperature ≥ 38.0°C or axillary temperature ≥ 37.4°C) or acute illness on the day of inclusion.

Ages: 42 Days to 56 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety of DTacP-IPV//PRP~T combined vaccine | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- New Delhi, India

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com